CLINICAL TRIAL: NCT06185543
Title: A Phase 2, Randomized, Prospective Double-Blind, Single-Center, Placebo-controlled Study to Evaluate Safety, Tolerability, Target Engagement, and Efficacy of PrimeC in Patients With Mild to Moderate Alzheimer's Disease (AD)
Brief Title: A Phase 2, Randomized, Prospective Double-Blind, Single-Center, Placebo-controlled Study to Evaluate Safety, Tolerability, Target Engagement, and Efficacy of PrimeC in Patients With Mild to Moderate Alzheimer's Disease.
Acronym: RoAD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroSense Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NST-AD-001
Record Dates: First submitted 2023-11-28; First posted 2023-12-29 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PrimeC (Active Comparator): 2 tablets of PrimeC administered twice daily (4 tablets a day), total daily dose of 1360 mg ciprofloxacin and 136 mg celecoxib orally.
  Interventions: Drug: PrimeC
- Placebo (Placebo Comparator): 2 tablets of Placebo administered twice daily (4 tablets a day). Placebo tablets are matched in size, color and taste.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PrimeC — Ciprofloxacin and celecoxib combination extended release formulation
  Arms: PrimeC
Drug: Placebo — Placebo matches active drug in size, color and taste
  Arms: Placebo

SUMMARY:
20 subjects with mild to moderate AD will be enrolled in the study and randomized at a 1:1 ratio to receive the study drug or placebo tablets, respectively. All subjects will be administered the drug/placebo twice daily (BID), two tablets each time, for 52 weeks.

Subjects will be allowed to receive standard of care (SOC) treatment of approved products or their combination. Subjects will be evaluated every 3 months for safety and tolerability.

DETAILED DESCRIPTION:
This is a Phase II, Randomized, Single-center, Prospective, Double-Blind, Placebo-Controlled Study, to evaluate Safety, Tolerability, target engagement and efficacy of PrimeC in subjects with mild to moderate AD. Subjects who meet the inclusion criteria and none of the exclusion criteria and who provide a signed Informed Consent will be enrolled in the study.

20 subjects with mild to moderate AD will be enrolled in the study and randomized at a 1:1 ratio to receive the study drug or placebo tablets, respectively. All subjects will be administered the drug/placebo twice daily (BID), two tablets each time, for 52 weeks.

Subjects will be allowed to receive standard of care (SOC) treatment of approved products or their combination (rivastigmine, donepezil, galantamine, memantine, donezepil, aducanumab, and lecanemab).

Subjects will be evaluated every 3 months for safety and tolerability (adverse events, safety laboratory, vital signs, ECG, withdrawal rates and reasons). Subjects will be evaluated for efficacy at baseline and after 12 months for CSF biomarkers and clinical outcomes (CDR, ADAS COG 14, ADCS-iADL, MMSE), for blood biomarkers at baseline, 6 and 12 months, and for C-SSRS every 3 months. A remote follow up (via phone call) will be conducted 1 month after baseline visit in order to confirm investigational drug compliance according to the protocol and potential AEs.

Adverse events (AEs) including any death, will be recorded throughout the study.

During the study, the sponsor, the PI, the outcome assessor, the subjects and all staff involved in the collection and recording of the clinical and laboratory data will be blinded to the treatment assignment. In addition, all aspects of data management and clean-up will be done using blinded datasets.

Following completion of 12 months of treatment, data lock will be performed, and data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF) and their ability to consent was estimated by an independent Neurologist or Geriatrist.
2. Males or females between the ages of 55 and 85 years of age, inclusive
3. Diagnosis of probable AD with evidence of the AD pathophysiological process according to the diagnostic criteria of the National Institute on Aging and Alzheimer's Association
4. AD patients with a score of 18 to 24 on MMSE at screening.
5. Subjects may be treated in parallel with rivastigmine, donepezil, galantamine, memantine, donezepil, aducanumab, and lecanemab or their combination. For rivastigmine, donepezil, galantamine, memantine, donezepil - 30 days of stable use prior to enrollment is required. For aducanumab and lecanemab - 3 months of stable use prior to enrollment is required.
6. 18 < BMI < 30
7. Patients who have a caregiver - the caregiver shall be in contact with the patient at least 10 hours per week, and can attend all visits with the patient, report on the subject's status and verify compliance with all study requirements.
8. CT or MRI available within 12 months before the enrolment to the study devoid of any structural finding which could explain the cognitive impairment, except for brain atrophy or white matter hyperintensities which can be observed in AD patients.
9. CT or MRI available within 3 months before the lumbar puncture.
10. Presence of pTau 181 in CSF at screening
11. Female with no childbearing potential (at least 1 year postmenopausal or surgical contraception)

Exclusion Criteria:

1. Any significant neurologic or medical disorders other than AD, which might be the cause of the existing cognitive deficit, such as: other neurodegenerative disease, Hydrocephalus including NPH, seizures, Huntington's disease, Amyotrophic lateral sclerosis, multiple sclerosis, systemic lupus erythematosus, progressive supranuclear palsy, neurosyphilis, HIV, learning disability, intellectual disability, hypoxic cerebral damage, relevant neoplasm, toxic exposure, or any significant medical conditions that, in the opinion of the PI would endanger the health and wellbeing of the participant.
2. Stroke or Transient Ischemic Attack (TIA) within 6 months of screening visit.
3. History of severe head trauma with documented loss of consciousness or with radiological findings associated with the injury, leading to other neurological deficits.
4. Any contraindication to conduct lumber puncture.
5. Major depressive disorder according to DSM-V criteria requiring hospitalization within the previous 90 days before screening.
6. Suicidal ideation and behavior assessed by C-SSRS.
7. Serum B12 clinically significantly below the lower limit of normal at screening
8. Patients with history or current evidence of clinical significant peripheral neuropathy. The severity of the peripheral neuropathy will be determined by the investigator.
9. Patients who take tizanidine
10. Patients with history or current clinically significant of psychiatric disorders (e.g., anxiety, depression, delirium) occurring within the last two years, which required the subject to be hospitalized.
11. Patients with known history of myasthenia gravis or myasthenic syndrome
12. No psychotropics can be started during the trial except for short acting hypnotics for sleep and or low potency neuroleptics for agitation.
13. If the patient is taking antipsychotic, antidepressant, antianxiety or any other psychotropic before enrollment to the study there was no dose change 30 days before enrollment.
14. A past history of adverse reaction/hypersensitivity to either NSAIDs, celecoxib or fluoroquinolones, ciprofloxacin and / or to the non-active components of PrimeC: Microcrystalline cellulose Avicel, Povidone K-30, Sodium lauryl sulphate, Hydroxy propyl methyl cellulose, Microcrystalline cellulose, Colloidal Silicon Dioxide, Magnesium Stearate, and Opadry Blue.
15. Any known clinically significant abnormal gastric mucosal erosion, ulcer or tumor or/and GI disorder and/or bariatric surgery
16. Known history of clinically significant impairment of renal function (eGFR < 60)
17. Known or suspected symptomatic congestive heart and/or coronary heart disease, previous history of myocardial infarction, CABG, uncontrolled arterial hypertension, or rhythm abnormalities requiring permanent treatment
18. Known history of QT/QTc prolongation, Torsade de pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT syndrome) and the use of concomitant medications that prolong the QT/QTc interval.
19. Patients with known aortic aneurysms and heart valve regurgitation/incompetence.
20. Known or suspected diagnosis or family history of epilepsy in first degree relatives.
21. Known predisposition to tendinitis.
22. Known Impaired hepatic function.
23. Known or suspected to be a poor CYP2C9 metabolizer who also uses pharmacologic agents (prescription or over-the-counter) or herbal products known or suspected to induce or inhibit CYP2C9 within 30 days before enrollment.
24. Presence at screening of any medically significant cardiac, pulmonary, musculoskeletal, or psychiatric illness that might interfere with the subject's ability to comply with study procedures or that might confound the interpretation of clinical safety data, including, but not limited to:

    1. Mean systolic blood pressure >160 mm Hg and/or mean diastolic blood pressure >100 mm Hg (measurements taken after a few minutes rest) that persist on 3 successive measurements taken at least 2 minutes apart
    2. NYHA Class II or greater congestive heart failure
    3. Chronic obstructive pulmonary disease or asthma requiring daily use of bronchodilator medications
    4. Uncontrolled diabetes mellitus
25. Subject who is treated with chronic aspirin or NSAIDs and is at risk if stopped. Clopidogrel is allowed and can replace Aspirin.
26. Any contraindication for ciprofloxacin and celecoxib according to the current prescribing information.
27. Any impairment or social circumstance that, in the opinion of the Investigator, would render the subject not suitable to participate in the study.
28. Subject, or subject's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
29. Subject is participating in (or plans to participate in) any other investigational drug trial or plans to be exposed to any other investigational agent, device and/or procedure, from 30 days prior to Screening through study completion.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-11-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
To assess safety and tolerability of PrimeC in mild to moderate AD patients (change from baseline to 12 months) | 12 months
  * Incidence and severity of treatment-emergent adverse events (TEAEs)
  * Number (%) of subjects who discontinued treatment prematurely
  * Number (%) of subjects who discontinued treatment prematurely due to AEs
  * Number (%) of subjects with clinically significant abnormal laboratory values following treatment

SECONDARY OUTCOMES:
To assess the effect of PrimeC on cognitive functioning and activities of daily living in mild to moderate AD patients (change from baseline to 12 months) | 12 months
  The mean difference from baseline to 12 months between PrimeC and Placebo in Clinical Dementia Rating Scale (CDR)
To assess the effect of PrimeC on cognitive functioning and activities of daily living in mild to moderate AD patients (change from baseline to 12 months) | 12 months
  • The mean difference from baseline to 12 months between PrimeC and Placebo in the 13-item Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog 14)
To assess the effect of PrimeC on cognitive functioning and activities of daily living in mild to moderate AD patients (change from baseline to 12 months) | 12 months
  • The mean difference from baseline to 12 months between PrimeC and Placebo in the Alzheimer´s Disease Cooperative Study Activities of Daily Living Inventory Instrumental Items (ADCS-iADL)
To assess the effect of PrimeC on cognitive functioning and activities of daily living in mild to moderate AD patients (change from baseline to 12 months) | 12 months
  • The mean difference from baseline to 12 months between PrimeC and Placebo in the Mini-Mental State Examination (MMSE)

OTHER OUTCOMES:
Exploratory | 12 months
  : To explore the effect of PrimeC on AD specific biofluid (plasma and CSF) markers, AD-related hallmarks, and target engagement markers in mild to moderate AD patients (change from baseline to 12 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided